CLINICAL TRIAL: NCT01614587
Title: Do Patients With Early Post Operative Recurrence of Pelvic Organ Prolapse Have a Genetic Predisposition?
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Collaborators: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: R11-10-004
Record Dates: First submitted 2012-05-31; First posted 2012-06-08 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; recurrence of pelvic organ prolapse; genetic predisposition; SNP microarray analysis; pelvic floor; genetic factors; adequate prolapse repair; polymorphisms; surgical failure; reoperation; DNA; buccal swabs; TaqMan SNP allelic discriminiation assays; duplex real-time PCR; genome-wide SNP microarrays; next-generation sequencing
MeSH Terms: conditions — Pelvic Organ Prolapse; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA obtained from a buccal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases: 1. Early, unexplained recurrence (within six months of procedure) after Sacrocolpopexy
  2. The recurrence required treatment (surgery or pessary)
- Controls: 1. Sacrocolpopexy during the same period
  2. No recurrence, no reoperation, no retreatment to date (minimum of 12 months from surgery)

SUMMARY:
The objective is to explore the genetic predisposition to early pelvic organ prolapse after adequate surgical repair by exploring the association between pelvic organ prolapse recurrences and certain polymorphisms.

DETAILED DESCRIPTION:
Pelvic organ prolapse develops as a result of a loss of support provided by the muscles and fascia that constitute the pelvic floor. Several recent population studies have estimated the prevalence of pelvic organ prolapse at between 10% and 30%. One in nine women will undergo surgery for these disorders in her lifetime and of these, one third will undergo repeated surgeries. The correction of pelvic organ protrusion is aimed at restoring the pelvic floor functional status and ultimately improving the patients quality of life. There are a few studies that have explored the genetic predisposition to developing pelvic organ prolapse but none so far looks at genetic factors involved in prolapse recurrence after adequate prolapse repair. There are two groups of women: women who underwent adequate repair of their prolapse and had an unexplained early recurrence. And a second control group of women who underwent the same prolapse repair procedure and had no further prolapse recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Cases: early, unexplained recurrence (within 6 months of procedure) after sacrocolpopexy), the recurrence required treatment (surgery or pessary) Controls: sacrocolpopexy during the same period, no recurrence, no reoperation, no retreatment to date (minimum of 12 months from surgery)

Exclusion Criteria:

* Obvious surgical technical failure
* Use of other graft material than polypropylene mesh
* Planned two staged operation
* Contraindications to surgery based on existing medical conditions
* Pregnancy
* Desire for pregnancy in the future

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women suffering from pelvic organ prolapse
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
SNP microarray analysis from recurrent prolapse subjects and controls | 12 months post-operative, DNA will be collected
  DNA will be evaluated by a variety of methods. For example, candidate polymorphisms may be evaluated using TaqMan SNP allelic discrimination assays which are based upon duplex real-time PCR. In addition, genome-wide SNP microarrays may be employed in order to perform a whole genome association study. Additional analysis such as DNA resequencing may also be required in order to identify causative polymorphisms linked to the newly associated SNPs. Other methods of DNA analysis such as next-generation sequencing may also be warranted.

SECONDARY OUTCOMES:
Compare all peri-operative characteristics and demographics between groups | 12 months post-operative
  Perioperative data will include: age, date of surgery, repeat procedure or treatment, procedure and mesh used, mesh related complications, early post-operative complications. Descriptive statistics will be derived for the entire group. The two subgroups (case and control) will then be compared using: Student t test, Fisher exact test, and Wilcoxon rank-sum test for continuous, nonparametric categorical and nonparametric ordinal variables, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Scott, MD, Principal Investigator — Reproductive Medicine Associates; Patrick Culligan, MD, Principal Investigator — Atlantic Health System; Charbel Salamon, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health System, Morristown, New Jersey, United States

REFERENCES:
- [Derived] St Louis S, Scott R, Lewis C, Salamon C, Pagnillo J, Treff N, Taylor D, Culligan P. Genetic Mutation that May Contribute to Failure of Prolapse Surgery in White Women: A Case-Control Study. J Minim Invasive Gynecol. 2016 Jul-Aug;23(5):726-30. doi: 10.1016/j.jmig.2016.02.019. Epub 2016 Mar 2. PMID 26944198